CLINICAL TRIAL: NCT02461940
Title: A Randomized Controlled Trial of an STI/HIV/AIDS Prevention Intervention for Adolescents Attending a Public STI Clinic in Singapore
Brief Title: STI/HIV Prevention Intervention for Adolescents in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); National Skin Centre, Singapore (Other)
Responsible Party: Principal Investigator, Wong Mee Lian, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMRC/1188/2008
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Sexually Transmitted Infections
Keywords: Sexual behavior; condom use; secondary abstinence
MeSH Terms: conditions — Sexually Transmitted Diseases; Sexual Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): The control group will receive the standard care provided by the STI clinic.
- Adolescent Behavioral intervention (Active Comparator): Participants allocated to the intervention arm receive 4 on-site personalised counselling and 2 phone/online sessions over a 12-month period, targeting individual, relational, sociocultural and environmental factors pertaining to the acquisition of STI/HIV.
  Interventions: Behavioral: Adolescent Behavioral Intervention

INTERVENTIONS:
Behavioral: Adolescent Behavioral Intervention — Session 1 focuses on STI/HIV education and self-reflection. Session 2 aims to increase the awareness of STI/HIV preventive strategies by instilling condom use and negotiation skills. Motivational Interviewing is used during the behavioural counselling. Session 3 reviews the goal on safer sex set by the participant and examines the successful strategies on safer sex and identifies triggers for relapse. Success stories are shared to renew their motivation. Session 4 reinforces the progress of the participant by recapitulating the knowledge and motivation explored in previous sessions. The online sessions, by phone/SMS/Whatsapp are conducted 2 months after the second and third sessions to find out if they face any difficulties and to reinforce prevention information covered previously.
  Arms: Adolescent Behavioral intervention

SUMMARY:
A randomized controlled trial conducted on 688 sexually experienced adolescents, with 337 participants assigned to the routine program, and 351 to the new intervention developed from an assessment of their needs. All participants will complete a self-administered questionnaire and an interview on their knowledge of sexually transmitted infections (STIs)/Human Immunodeficiency Virus (HIV), self-efficacy, skills in negotiating for sexual abstinence or condom use, and sexual behaviors at baseline and at 6- and 12-months' post- intervention. All will be tested for STIs. Participants in the intervention group will receive 4 individual counseling sessions on STIs/HIV knowledge, life skills, secondary abstinence, safer sex and healthy relationships over 1 year. They will also be referred to counselors for proactive social and emotional support delivered through electronic media and other means. The control group will receive the usual counseling session at first and follow-up clinic visit.

DETAILED DESCRIPTION:
The reasons for conducting this study in a clinical setting is threefold.

1. This is group of adolescents that has a high risk for transmitting STIs to the community. Prior to this intervention, the investigators did a preliminary study and found a high number of sex partners (median: 4, range: 1-25) and high prevalence of unprotected sex (90%) and STIs (60%) in this group. Other factors in this group that facilitate the transmission of STIs is that 36% continued to engage in unprotected sex and half of the boys (49%) and three quarters of the girls (77%) delayed seeking treatment for more than a week after experiencing symptoms of STIs. The rate at which STIs spread in a population depends upon the average number of new cases of infection generated by an infected person (the basic or case reproduction ratio (Ro). This ratio, in turn, depends upon the efficiency of transmission, (b), the mean rate of change of sexual partners (c), and the average duration of infectiousness (D) as expressed in the form: Ro=b*c*D. Given their high number of sex partners and the long duration of infectiousness owing to their delay in seeking treatment, they would form an important group for spreading STIs to the general population.
2. The investigators are able to adopt a rigorous study design, that is, a randomized controlled trial in a clinical setting to evaluate the efficacy of the intervention, and validate self-reported behaviors with laboratory tests for STIs. In contrast, it is less feasible to conduct the study in schools presently because of the sensitivity of the topic, conservative attitudes of parents and possible biases of self-reported sexual behavior in schools. School-based interventions will also exclude school drop outs, who were found in this ongoing study, to be significantly, more likely to engage in sexual activity.
3. The investigators have conducted needs assessment of this group and this would help in developing interventions specifically for them. For instance, the investigators found that both males and females lack the confidence of using condoms correctly. The investigators incorporated a session on instilling skills for condom use in our intervention.

ELIGIBILITY:
Inclusion Criteria:

* Singaporean citizens or permanent residents
* Sexually active for the past 1 year
* Heterosexual
* Attending the clinic for the first time
* Able to commit for one year in Singapore

Exclusion Criteria:

* Involved in criminal investigation

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 688 (Actual)
Dates: Start 2009-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Consistent condom use | 12 months
  This is assessed by: "Have you or your partner ever used a condom for vaginal sex in the last 6 months?" in the survey. Participants who gave the answer as 'Yes, always' are categorised as having consistent condom usage; whereas those who gave the answer as "Yes, sometimes", "No, not at all" and "Can't remember" are categorised as having inconsistent condom use.
Secondary abstinence | 12 months
  This is assessed by: "How many times did you have vaginal sex in the last 6 months?"
STI incidence | 12 months
  Defined as having a positive laboratory test result for a new episode of chlamydia, gonorrhoea, herpes, syphilis or HIV infection at either the 6-month or the 12-month assessment. Both gonorrhoea and chlamydia are detected by testing the urine specimens using Cobas Amplicor Polymerase Chain Reaction (PCR) assay. Type-specific serological tests (TSSTs) based on glycoprotein gG-1 and/or gG-2 are used to identify patients with genital herpes. Syphilis is screened using Enzyme Immunoassay (EIA) treponemal test. HIV rapid test is performed using the Determine HIV-1/HIV-2 (Abbott) rapid test kit, where results are available in 20 minutes. For those who do not want to wait may opt for the EIA test for HIV infection.
Number of sexual partners | 12 months
  This is is assessed by "How many persons did you have sex with in the last 6 months?"
Consistent condom use | 6 months
  This is assessed by: "Have you or your partner ever used a condom for vaginal sex in the last 6 months?" in the survey. Participants who gave the answer as 'Yes, always' are categorised as having consistent condom usage; whereas those who gave the answer as "Yes, sometimes", "No, not at all" and "Can't remember" are categorised as having inconsistent condom use.
Secondary abstinence | 6 months
  This is assessed by: "How many times did you have vaginal sex in the last 6 months?"
STI incidence | 6 months
  Defined as having a positive laboratory test result for a new episode of chlamydia, gonorrhoea, herpes, syphilis or HIV infection at either the 6-month or the 12-month assessment. Both gonorrhoea and chlamydia are detected by testing the urine specimens using Cobas Amplicor Polymerase Chain Reaction (PCR) assay. Type-specific serological tests (TSSTs) based on glycoprotein gG-1 and/or gG-2 are used to identify patients with genital herpes. Syphilis is screened using Enzyme Immunoassay (EIA) treponemal test. HIV rapid test is performed using the Determine HIV-1/HIV-2 (Abbott) rapid test kit, where results are available in 20 minutes. For those who do not want to wait may opt for the EIA test for HIV infection.
Number of sexual partners | 6 months
  This is assessed by "How many persons did you have sex with in the last 6 months?"

SECONDARY OUTCOMES:
Success in stopping pressured sex | 12 months
  This is assessed by: "If a boy/ girl puts pressure on you to be involved sexually and you don't want to be involved, how often do you succeed in stopping it?"
Confidence in using condoms correctly | 12 months
  This is assessed by "How confident are you that you are using the condom correctly?" and rated on a scale ranging from "not confident at all" to "very confident"
Confidence in negotiating for condom use | 12 months
  This is evaluated by "How confident are you that you are able to persuade your boyfriend/girlfriend to use condom?"
Success in stopping pressured sex | 6 months
  This is assessed by: "If a boy/ girl puts pressure on you to be involved sexually and you don't want to be involved, how often do you succeed in stopping it?"
Confidence in using condoms correctly | 6 months
  This is assessed by "How confident are you that you are using the condom correctly?" and rated on a scale ranging from "not confident at all" to "very confident"
Confidence in negotiating for condom use | 6 months
  This is evaluated by "How confident are you that you are able to persuade your boyfriend/girlfriend to use condom?"

CONTACTS AND LOCATIONS:
Overall Officials: Mee-Lian Wong, MPH, MD, Principal Investigator — National University of Singapore

REFERENCES:
- [Background] Wong ML, Chan RK, Koh D, Tan HH, Lim FS, Emmanuel S, Bishop G. Premarital sexual intercourse among adolescents in an Asian country: multilevel ecological factors. Pediatrics. 2009 Jul;124(1):e44-52. doi: 10.1542/peds.2008-2954. PMID 19564268
- [Background] Wong ML, Chan RK, Tan HH, Sen P, Chio M, Koh D. Gender differences in partner influences and barriers to condom use among heterosexual adolescents attending a public sexually transmitted infection clinic in Singapore. J Pediatr. 2013 Mar;162(3):574-80. doi: 10.1016/j.jpeds.2012.08.010. Epub 2012 Sep 20. PMID 23000347
- [Background] Kipke MD, Boyer C, Hein K. An evaluation of an AIDS risk reduction education and skills training (ARREST) program. J Adolesc Health. 1993 Nov;14(7):533-9. doi: 10.1016/1054-139x(93)90136-d. PMID 8312288
- [Background] Sen P, Chio MT, Tan HH, Chan RK. Rising trends of STIs and HIV infection in Singapore-- a review of epidemiology over the last 10 years (1994 to 2003). Ann Acad Med Singap. 2006 Apr;35(4):229-35. PMID 16710492
- [Background] Wong ML, Sen P, Wong CM, Tjahjadi S, Govender M, Koh TT, Yusof Z, Chew L, Tan A, K V. Human immunodeficiency virus (HIV) prevention education in Singapore: challenges for the future. Ann Acad Med Singap. 2012 Dec;41(12):602-9. PMID 23303119
- [Derived] Ng JYS, Chan RKW, Chio MT, Lim RBT, Koh D, Wong ML. An Abstinence and Safer Sex Intervention for Adolescents Attending the Public Sexually Transmitted Infection Clinic in Singapore. J Adolesc Health. 2018 Jun;62(6):737-746. doi: 10.1016/j.jadohealth.2017.12.014. Epub 2018 Apr 13. PMID 29661642